CLINICAL TRIAL: NCT04068480
Title: Study of Esophageal and Gastric Diseases With Robotically Controlled Magnetic Capsule Endoscopy
Brief Title: Esophageal and Gastric Diseases With Robotically Controlled Magnetic Capsule Endoscopy
Acronym: MACEOES
Status: Recruiting | Type: Observational
Sponsor: Bács-Kiskun County Teaching Hospital (Other)
Responsible Party: Principal Investigator, László Madácsy Md, PhD, Clinical Professor, Bács-Kiskun County Teaching Hospital
Other Study IDs: BacsKiskunCTH
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Video Capsule Endoscopy; Esophageal Diseases
Keywords: capsule endoscopy; magnetically assisted capsule endoscopy; MCCE; Esophagus; non-invasive endoscopy
MeSH Terms: conditions — Esophageal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Capsule endoscopy patients: Patients swallowed the capsules in left lateral position, leaning on their left forearms and elbows, while we were positioning the magnet tightly against their backs. With the magnetic field vector X,Y,Z axis 180, -90 and 90, respectively. After swallowing the capsules with a small amount of water, they remained in this left lateral decubitus position.

SUMMARY:
Magnetically controlled capsule endoscopy (MCCE) is an outstanding opportunity for the painless endoscopic screening of the esophagus and stomach before small bowel examiantion. Further improvement in patients positioning might increase the esophageal transit time of the capsule endoscope and could improve the sensitivity and specificity of the esophageal MCCE investigation. Our present study aimed to compare the visualization of the esophagus (especially the Z-line) with different capsule swallowing protocols.

DETAILED DESCRIPTION:
Magnetic controlled capsule endoscope (MCCE) systems have been developed over the last 10-15 years to examine the upper GI tract, particularly the stomach. The new Navicam MACE system consists of a magnetic capsule endoscope, an external control magnet, a data recording kit and a computer workstation. With the appropriate software, allows real-time tracking and monitoring of the capsule inside the body. This method may in the near future be an optimal non-invasive method for screening gastric cancer and Barrett's oesophagus in high-risk populations.

Esophagogastroduodenoscopy (EGD) is the gold standard diagnostic test, however it is very inconvenient for patients without sedation.

The aim of our present study was a feasibility study to evaluate the safety and efficacy of Ankon MCCE for the investigation of esophageal abnormalities in patients referred for small bowel capsule endoscopy in our endoscopy department, to develop and test a method to use MCCE for esophageal examination, and to analyze the visualization of esophageal mucosa with our newly developed capsule swallowing protocol and manual capsule maneuvering.

ELIGIBILITY:
Inclusion Criteria:

- patients referred for small bowel capsule endoscopy in any indication

Exclusion Criteria:

* known or suspected stricture in the GI tract
* previous surgery with bowel anastomosis
* swallowing complaints
* dementia
* implanted cardioverter defibrillator
* inability to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient who met the eligibility criteria and had MCCE examination with esophageal protocol.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-11-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Reflux esophagitis | 1 year
  Proportion and the severity of reflux (Los Angeles classification) comparing to gastroscopy
Diseases | 1 year
  Proportion of other disorders of oesophagus and stomach comparing to gastroscopy
Stomach examination | 1 year
  Analyze the visualisation of gastric mucosa with MACE system

SECONDARY OUTCOMES:
Restrain time | 1 year
  Analysing the correlation with MCCE system between esophageal transit time and diagnostic yield.
Cleanliness | 1 year
  Analysis of stomach preparation with a special software concerning the percentage of clean and covered areas.

CONTACTS AND LOCATIONS:
Overall Officials: László Madácsy, Prof., Principal Investigator — Bács-Kiskun County Teaching Hospital
Locations (1):
- Endo-Kapszula Privat Medical Cenbter, Székesfehérvár, --None---, Hungary